CLINICAL TRIAL: NCT00324324
Title: Randomized, Double Blinded, Placebo-Controlled Trial of Antibacterial Prophylaxis for the Prevention of Bacterial Infections in the Post-Engraftment Phase After Allogeneic Hematopoeitic Stem Cell Transplantation
Brief Title: Moxifloxacin in Preventing Bacterial Infections in Patients Who Have Undergone Donor Stem Cell Transplant
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Joseph Bubalo, PharmD, OHSU Knight Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CDR0000472877; P30CA069533 (NIH); OHSU-TPI-02027-L (Other: Oregon Health and Science University); OHSU 0285 (Other: Oregon Health & Science University)
Record Dates: First submitted 2006-05-10; First posted 2006-05-11 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Breast Cancer; Chronic Myeloproliferative Disorders; Gestational Trophoblastic Tumor; Infection; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms; Neuroblastoma; Ovarian Cancer; Testicular Germ Cell Tumor
Keywords: infection; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); accelerated phase chronic myelogenous leukemia; adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; atypical chronic myeloid leukemia, BCR-ABL negative; blastic phase chronic myelogenous leukemia; chronic eosinophilic leukemia; primary myelofibrosis; chronic myelomonocytic leukemia; chronic neutrophilic leukemia; chronic phase chronic myelogenous leukemia; de novo myelodysplastic syndromes; disseminated neuroblastoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; myelodysplastic/myeloproliferative neoplasm, unclassifiable; nodal marginal zone B-cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; poor prognosis metastatic gestational trophoblastic tumor; previously treated myelodysplastic syndromes; recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; recurrent adult Burkitt lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent mycosis fungoides/Sezary syndrome; recurrent neuroblastoma; recurrent ovarian epithelial cancer; recurrent ovarian germ cell tumor; recurrent small lymphocytic lymphoma; recurrent malignant testicular germ cell tumor; refractory chronic lymphocytic leukemia; refractory hairy cell leukemia; refractory multiple myeloma; relapsing chronic myelogenous leukemia; secondary acute myeloid leukemia; secondary myelodysplastic syndromes; splenic marginal zone lymphoma; stage I multiple myeloma; stage II multiple myeloma; stage II ovarian epithelial cancer; stage III adult Burkitt lymphoma; stage III adult Hodgkin lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III chronic lymphocytic leukemia; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III multiple myeloma; stage III ovarian epithelial cancer; stage III small lymphocytic lymphoma; stage III malignant testicular germ cell tumor; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV adult Burkitt lymphoma; stage IV adult Hodgkin lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV breast cancer; stage IV chronic lymphocytic leukemia; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV ovarian epithelial cancer; stage IV small lymphocytic lymphoma
MeSH Terms: conditions — Breast Neoplasms; Myeloproliferative Disorders; Gestational Trophoblastic Disease; Infections; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Neuroblastoma; Ovarian Neoplasms; Testicular Germ Cell Tumor; Congenital Abnormalities; Leukemia, Myeloid, Accelerated Phase; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Pdgfra-Associated Chronic Eosinophilic Leukemia; Primary Myelofibrosis; Leukemia, Myelomonocytic, Chronic; Leukemia, Neutrophilic, Chronic; Leukemia, Myeloid, Chronic-Phase; Lymphoma, B-Cell, Marginal Zone; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Burkitt Lymphoma; Hodgkin Disease; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Carcinoma, Ovarian Epithelial; Leukemia, Lymphocytic, Chronic, B-Cell; Testicular Neoplasms; Leukemia, Hairy Cell | interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- moxifloxacin hydrochloride (Active Comparator): Moxifloxacin 400 mg capsule orally once a day through D+100 after bone marrow transplant, then discontinue
  Interventions: Drug: moxifloxacin hydrochloride
- Sugar pill (Placebo Comparator): Placebo 1 capsule orally once a day through D+100 after bone marrow transplant, then discontinue
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: moxifloxacin hydrochloride — Moxifloxacin/Placebo 400 mg capsule orally once a day through D+100 after bone marrow transplant, then discontinue
  Arms: moxifloxacin hydrochloride
Drug: Placebo — Moxifloxacin/Placebo 400 mg capsule orally once a day through D+100 after bone marrow transplant, then discontinue
  Arms: Sugar pill

SUMMARY:
RATIONALE: A donor stem cell transplant can lower the body's immune system, making it difficult to fight off infection. Giving antibiotics, such as moxifloxacin, may help prevent bacterial infections in patients who have recently undergone donor stem cell transplant. It is not yet known whether moxifloxacin is more effective than a placebo in preventing bacterial infections in patients who have recently undergone donor stem cell transplant.

PURPOSE: This randomized phase III trial is studying moxifloxacin to see how well it works compared with a placebo in preventing bacterial infections in patients who have recently undergone donor stem cell transplant.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess the safety and tolerability of giving prophylactic moxifloxacin hydrochloride during the post-engraftment phase in patients who have undergone allogeneic stem cell transplantation. (Pilot study)
* Compare the efficacy, in terms of reducing the incidence of clinically and microbiologically documented bacterial infections, in patients who have undergone allogeneic stem cell transplantation treated with prophylactic moxifloxacin hydrochloride vs placebo during the post-engraftment phase. (Phase III)

Secondary

* Determine the incidence of clinically and microbiologically documented bacterial infections in these patients. (Pilot study)
* Assess the impact of moxifloxacin hydrochloride on the incidence of bacteremia in these patients. (Phase III)
* Compare the percentage of time on systemic antibiotics and days hospitalized in patients treated with these regimens. (Phase III)
* Compare the incidence of veno-occlusive disease of the liver in patients treated with these regimens. (Phase III)
* Compare the incidence and severity of graft-versus-host disease in patients treated with these regimens. (Phase III)
* Compare the infection-related mortality and overall mortality of patients treated with these regimens.

OUTLINE: This is a pilot study followed by a randomized, double-blind, placebo-controlled, multicenter phase III study. Patients are stratified according to gender and race (white vs. non-white). The first 20 patients are assigned to the pilot study.

Patients assigned to the pilot study receive oral moxifloxacin hydrochloride once daily beginning after neutrophil recovery (ANC > 1,500/mm³) from allogeneic stem cell transplantation (ASCT) and continuing until day 100 post-transplantation in the absence of disease progression or unacceptable toxicity. Subsequent patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral moxifloxacin hydrochloride once daily beginning after neutrophil recovery (ANC > 1,500/mm³) from ASCT and continuing until day 100 post-transplantation.
* Arm II: Patients receive oral placebo once daily beginning after neutrophil recovery (ANC > 1,500/mm³) from ASCT and continuing until day 100 post-transplantation.

In both arms, treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at day 120 post-transplantation.

PROJECTED ACCRUAL: A total of 240 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Must be planning to undergo or have completed allogeneic stem cell transplantation (ASCT)

  * Must not be undergoing a nonmyeloablative ASCT
* Must not require antibiotic prophylaxis against bacterial pathogens during the post-engraftment phase as per ASCT protocol
* No known colonization with an antimicrobial-resistant organism normally sensitive to quinolones that is known to increase infection incidence (i.e., ciprofloxacin-resistant Pseudomonas not allowed; vancomycin-resistant Enterococcus and methicillin-resistant Staphylococcus aureus allowed)

PATIENT CHARACTERISTICS:

* Life expectancy ≥ 100 days
* Not pregnant or nursing
* Fertile patients must use effective contraception
* Negative pregnancy test
* No known hypersensitivity to fluoroquinolones
* No prolonged QTc interval on EKG (i.e., QTc > 440 milliseconds)
* No uncontrolled hypokalemia

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No concurrent class IA (e.g., quinidine or procainamide) or class III (e.g., amiodarone or sotalol) antiarrhythmics
* No concurrent intravenous antibiotics for pre-enrollment infections except vancomycin, linezolid, dalfopristin, or quinupristin (Synercid®)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2006-05; Primary Completion 2007-04 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | 1 to 120 days post bone marrow transplant

SECONDARY OUTCOMES:
Incidence of bacteremia | 1 to 120 days post bone marrow transplant
Incidence and severity of graft-versus-host disease | 1 to 120 days post bone marrow transplant
Infection-related mortality | 1 to 120 days post bone marrow transplant
Overall mortality | 1 to 120 days post bone marrow transplant

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Bubalo, PharmD, BCPS, BCOP, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- Knight Cancer Institute at Oregon Health and Science University, Portland, Oregon, United States

REFERENCES:
- [Result] Bubalo JS, Leis JF, Curtin PT, et al.: A randomized, double-blinded, pilot trial of aprepitant added to standard antiemetics during conditioning therapy for hematopoietic stem cell transplant (HSCT). [Abstract] J Clin Oncol 25 (Suppl 18): A-9112, 520s, 2007.